CLINICAL TRIAL: NCT01354678
Title: Phase 1 Study to Evaluate the Efficacy and Safety of Intramyocardial Multiple Precision Injection of Bone Marrow Mononuclear Cells in Myocardial Ischemia
Brief Title: Intramyocardial Multiple Precision Injection of Bone Marrow Mononuclear Cells in Myocardial Ischemia
Acronym: IMPI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to inefficacy of the tested method
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMPI-1
Record Dates: First submitted 2011-05-13; First posted 2011-05-17 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure
Keywords: heart failure; bone marrow mononuclear cells
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group of bone marrow cell therapy (Active Comparator)
  Interventions: Procedure: NOGA XP Cardiac Navigation System
- group of sham therapy (Sham Comparator)
  Interventions: Procedure: NOGA XP Cardiac Navigation System

INTERVENTIONS:
Procedure: NOGA XP Cardiac Navigation System — Intramyocardial multiple precision injection of bone marrow mononuclear cells
  Other Names: Cordis Corporation's Biologics Delivery Systems
  Arms: group of bone marrow cell therapy
Procedure: NOGA XP Cardiac Navigation System — Intramyocardial multiple precision injection with placebo
  Other Names: Cordis Corporation's Biologics Delivery Systems
  Arms: group of sham therapy

SUMMARY:
Randomised placebo-controlled study of efficiency and safety of bone marrow mononuclear cells transplantation by intramyocardial multiple precision injection in ischemic heart failure patients.

DETAILED DESCRIPTION:
The increase of prevalence of heart failure in human population requires to develop new and effective methods of treatment. One of them is stem cells transplantation into a myocardial tissue, which cause the improvement of contractility, myocardial remodelling after myocardial infarction (MI), dilated cardiomyopathy, etc. Use of autologous stem cells does not require of immunosuppressive therapy and does not correlate with some ethical problems. Clinical application of mesenchymal stem cells always requires a step of culturing, which is associated with increased risk of contamination Therefore haemopoietic stem cells, endothelial progenitor cells or mononuclear bone marrow cells are often used to be transplant for treatment of heart failure (HF) patients.Using NOGA XP Cardiac Navigation System improves specificity of transplantations, that is decisive.

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary artery disease (CAD) and HF II-III NYHA class
* MI more than 6 months before the study
* LVEF less than 35%
* absence of indication to coronary revascularization
* optimal pharmacological therapy no less than 8 weeks
* heart transplantation is contraindicated
* patients with implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D)
* patients giving informed consent

Exclusion Criteria:

* acute coronary syndrome
* coronary revascularization less than 6 months
* patients requiring surgical correction of post-MI aneurism
* LV wall thickness less than 5 mm in site of possible injection
* patients with CRT implanted within 3 month before cells injection
* clinically significant associated diseases

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in global left ventricular ejection fraction and regional wall motion score index | 6 and12 months

SECONDARY OUTCOMES:
Incidence of the major adverse cardiac events | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eugene V Shlyakhto, Prof, Principal Investigator — Almazov Federal Heart, Blood and Endocrinology Centre
Locations (1):
- Almazov Federal National Medical Research Centre, Saint Petersburg, Russia